CLINICAL TRIAL: NCT07335289
Title: PrEP4U: Assessing the Effectiveness of Integrated Same-Day Lenacapavir Initiation and Follow-up Choice on PrEP Persistence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ruanne Barnabas, MBChB, MSc, DPhil., Chief, Division of Infectious Diseases, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025P002691
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: HIV Pre-exposure Prophylaxis Use
Keywords: HIV PrEP; Injectable PrEP; Lenacapavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PrEP Clinic (Active Comparator): The PrEP Clinic arm will be randomized to receive follow up at the clinic
  Interventions: Other: Follow up via standard clinic
- PrEP Choice (Experimental): The PrEP Choice arm allows participants to choose where they receive their follow up
  Interventions: Other: Choice of follow up

INTERVENTIONS:
Other: Choice of follow up — Randomization to either standard clinic follow up or choice of where follow up takes place
  Arms: PrEP Choice
Other: Follow up via standard clinic — Follow up will take place at the clinic where the first dose was administered.
  Arms: PrEP Clinic

SUMMARY:
PrEP4U is designed as a pragmatic, randomized implementation trial to test strategies that could directly inform real-world roll-out of lenacapavir. By integrating:

* Same-day initiation based on rapid HIV testing, and
* Choice of follow-up delivery location (home, community, or clinic) the study addresses two of the most pressing implementation questions for long-acting injectable PrEP.

The primary hypothesis is that giving participants choice in follow-up location will improve PrEP persistence compared to a clinic-only model. Secondary analyses will evaluate safety of rapid testing, acceptability, and participant costs. Exploratory analyses will assess HIV incidence and resistance.

Findings from PrEP4U will provide essential evidence to guide scalable, equitable, person-centered delivery models for lenacapavir PrEP in the U.S. and globally.

DETAILED DESCRIPTION:
Since the introduction of oral PrEP over a decade ago, more than 1.3 million HIV infections occur globally each year, far exceeding the UNAIDS 2030 target of < 335,000 cases. UNAIDS estimated that only 2.3 million people used PrEP in 2023, far below the target of 10 million by 2025. Oral PrEP persistence remains low, with many individuals discontinuing within 6-12 months. Factors contributing to low uptake and persistence include pill fatigue, stigma, access barriers, and medical mistrust. The gap is especially stark in sub-Saharan Africa and Latin America, where PrEP coverage lags behind epidemic burden.

The United States mirrors this global picture; despite broad access to healthcare, disparities in uptake and continuation persist along racial, ethnic, and gender lines. According to the CDC, in 2022 only 36% of individuals eligible for PrEP were prescribed it. Marked disparities exist: Black and Hispanic/Latino individuals and women represent a disproportionate share of new HIV diagnoses but a much smaller fraction of PrEP users. In Massachusetts, for example, Black and Hispanic/Latino individuals accounted for 35% and 31% of new HIV cases in 2022, yet only 7% and 12% of PrEP users in 2023, respectively. These disparities highlight ongoing barriers to access, stigma, and persistence.

Lenacapavir is a first-in-class HIV-1 capsid inhibitor with a novel mechanism of action and an exceptionally long half-life, enabling subcutaneous administration every 26 weeks. PURPOSE 1 and PURPOSE 2, large multicenter randomized clinical trials, established lenacapavir's efficacy for HIV prevention. In PURPOSE 2, a Phase 3 randomized trial of over 3,000 participants at risk for HIV infection, HIV incidence with lenacapavir was 0.10 per 100 person-years, compared to 0.93 per 100 person-years in the oral F/TDF arm and 2.37 per 100 person-years in the background incidence cohort. Lenacapavir reduced HIV incidence by 96% compared with background incidence and by 89% compared with oral PrEP. No major safety concerns were identified, though 1.2% discontinued due to injection-site reactions. These findings, published in the New England Journal of Medicine in 2025, demonstrated that twice-yearly lenacapavir is a highly effective PrEP agent.

Lenacapavir addresses key limitations of oral PrEP:

* Persistence challenges with daily oral adherence.
* Barriers to clinic attendance for frequent refills or injections.
* Stigma associated with oral PrEP use, which may be mitigated by less frequent, more discreet dosing.

Thus, lenacapavir has the potential to transform HIV prevention - if delivery strategies are optimized.

While clinical trials demonstrate efficacy, implementation science questions remain:

1. Same-day initiation: Oral PrEP initiation has successfully shifted to same-day models. However, injectable PrEP initiation has been complicated by requirements for multiple laboratory tests, delaying access. PURPOSE 1 and 2 used a combination of rapid HIV Ag/Ab, laboratory Ag/Ab, and quantitative RNA tests prior to injection. In real-world settings, RNA testing may be impractical and introduce delays. Rapid HIV testing, with confirmatory laboratory Ag/Ab tests pending, is a feasible approach aligned with WHO guidance. This balance enables timely initiation without undue barriers.
2. Follow-up and persistence: Lenacapavir's twice-yearly dosing reduces pill burden but raises questions of where and how injections are delivered. Relying on centralized hospital clinics may perpetuate barriers (transportation, stigma, scheduling). In contrast, home-based and community-based PrEP delivery have shown promise for improving persistence and acceptability.

Suffolk County, Massachusetts - home to central Boston - is designated a high-burden HIV area in the U.S. "Ending the HIV Epidemic" initiative, reporting 118 new HIV diagnoses in 2022. Despite broad health insurance coverage and a state-sponsored PrEP assistance program, PrEP uptake and persistence remain insufficient among Black, Hispanic/Latino, and female populations. PrEP4U will specifically recruit participants from these priority populations through community partner organizations, mobile van services, and clinical sites. The trial is designed to address equity gaps by testing models of care that reduce stigma, bring services closer to people, and incorporate patient choice.

ELIGIBILITY:
Inclusion Criteria:

* HIV negative
* Eligible for HIV PrEP per CDC guidelines
* Able and willing to provide informed consent
* Willing to receive injectable lenacapavir and adhere to study procedures
* Residing inMassachusetts with expected availability for 6-month follow-up

Exclusion Criteria:

* Known HIV infection at baseline
* Contraindication to lenacapavir injection (e.g., hypersensitivity, significant drug interactions)
* Pregnancy at baseline (participants who become pregnant during the trial may remain enrolled if they choose)
* Participation in another interventional HIV prevention study
* Any condition judged by the investigator to compromise safety or study integrity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
PrEP persistence at 6 months | 26 weeks
  Proportion of participants in the PrEP Choice arm versus the PrEP Clinic arm who successfully receive the second on-time injection

SECONDARY OUTCOMES:
Safety of same-day initiation based on rapid HIV testing | 26 weeks
  Proportion of individuals in whom rapid and laboratory Ag/Ab test results are consistent.
Acceptability of same-day initiation and follow-up models | 26 weeks
  Participant acceptability scores measured using structured surveys
Participant costs associated with PrEP delivery models | 26 weeks
  Average participant costs (financial and time) per injection visit in clinic versus community/home settings

OTHER OUTCOMES:
HIV Incidence by Study Arm | 26 weeks
  HIV incidence rate (per 100 person-years) by arm
Lenacapavir Resistance in HIV Seroconverters | 26 weeks
  Proportion of HIV infections with confirmed resistance mutations
Subgroup Analyses of Persistence | 26 weeks
  Identification of populations for whom differentiated delivery has the greatest impact

CONTACTS AND LOCATIONS:
Overall Officials: Ruanne V Barnabas, MBChB, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Sexual Health Clinic, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Interested parties may contact the central contact with requests for data. Data sets will be provided based on approval of request/concept by protocol team.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Once analysis of the study objectives is complete. Tentatively January 2027
Access Criteria: The protocol team will review all data requests. Upon approval of requests the data analyst will work with the requester to provide the data in an acceptable format, using a secure access link.